CLINICAL TRIAL: NCT00142233
Title: Double Blind Randomised Controlled Trial to Investigate the Efficacy of ANTOX (Vers) 1.2 and MGCT (Magnesiocard) for the Treatment of Hereditary Pancreatitis and Idiopathic Chronic Pancreatitis
Brief Title: EUROPAC-2 - Pain Treatment of Hereditary and Idiopathic Pancreatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EUROPAC-2
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Pancreatitis
Keywords: EUROPAC 2, ANTOX (vers)1.2, MGCT (Magnesiocard); Hereditary Pancreatitis; idiopathic chronic pancreatitis
MeSH Terms: conditions — Pancreatitis; Hereditary pancreatitis | interventions — Magnesium; Aspartic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ANTOX (vers.)1.2 (Experimental): Adults and children aged 10+ will take two ANTOX (vers)1.2 tablets three times per day. (Antioxidant treatment: daily: 300 μg organic selenium, 720 mg vitamin C, 228 mg vitamin E, 2880 mg methionine) plus two placebo Magnesiocard (2.5 mmol) tablets three times per day.
  Children aged five to nine years of age will take one ANTOX (vers)1.2 tablet three times daily (Antioxidant treatment: daily: 150 μg organic selenium, 360 mg vitamin C, 114 mg vitamin E, 1440 mg methionine) plus one placebo Magnesiocard (2.5 mmol) tablet three times a day.
  Interventions: Dietary Supplement: ANTOX (vers.)1.2; Other: Placebo Magnesiocard (2.5 mmol)
- Magnesium (Experimental): Adults and children aged 10+ will take two Magnesiocard (2.5 mmol) tablets three times per day (total dose: 15 mmol = 365 mg per day) plus two placebo ANTOX (vers)1.2 tablets three times a day.
  Children aged five to nine years of age will take one Magnesiocard (2.5 mmol) tablet three times a day (total dose: 7.5 mmol = 182 mg per day) plus one placebo ANTOX (vers)1.2 tablet three times a day.
  Interventions: Drug: Magnesium; Other: Placebo ANTOX (vers)1.2
- Placebo (Placebo Comparator): Adults and children aged 10+ will take two placebo ANTOX (vers)1.2 tablets three times a day, plus two placebo Magnesiocard (2.5 mmol) tablets three times per day.
  Children aged five to nine years of age will take one placebo ANTOX (vers)1.2 tablet three times a day, plus one placebo Magnesiocard (2.5 mmol) tablet three times per day.
  Interventions: Other: Placebo ANTOX (vers)1.2; Other: Placebo Magnesiocard (2.5 mmol)

INTERVENTIONS:
Dietary Supplement: ANTOX (vers.)1.2 — 300 µg organic selenium, 720 mg vitamin C, 228 mg vitamin E, 2880 mg methionine per day (for patients of 10 years and older)
  150 µg organic selenium, 360 mg vitamin C, 114 mg vitamin E, 1440 mg methionine per day (for patients aged between 5 and 9 years)
  Arms: ANTOX (vers.)1.2
Drug: Magnesium — 15 mmol per day (for patients of 10 years and older)
  7,5 mmol per day (for patients aged between 5 and 9 years)
  Other Names: Magnesiocard (MGCT)
  Arms: Magnesium
Other: Placebo ANTOX (vers)1.2 — Placebo ANTOX (vers)1.2
  Arms: Magnesium; Placebo
Other: Placebo Magnesiocard (2.5 mmol) — Placebo Magnesiocard (2.5 mmol)
  Arms: ANTOX (vers.)1.2; Placebo

SUMMARY:
This is a multi-centre randomised phase III, double blind, placebo controlled, parallel group, outpatient study in patients diagnosed with hereditary pancreatitis and idiopathic chronic pancreatitis.

The hypothesis to be tested is a 30% reduction in the number of days due to pancreatitis from 12.5 days per year to less than nine days per year under the treatment with magnesium or an antioxidant cocktail called ANTOX.

A total of 288 patients will be randomised to one of three treatment groups in order to compare pancreatic pain over a twelve month period.

DETAILED DESCRIPTION:
Title: EUROPAC 2 trial to investigate the efficacy of ANTOX (vers) 1.2 and MGCT (Magnesiocard) for the treatment of hereditary pancreatitis and idiopathic chronic pancreatitis

Study drug: ANTOX (vers) 1.2, MGCT (Magnesiocard)

Intended indication: Hereditary pancreatitis and idiopathic chronic pancreatitis

Study design: A multi-centre, double blind, and placebo-controlled, randomised, parallel group study

Patient population: Patients with hereditary pancreatitis or idiopathic chronic pancreatitis

Number of patients: Total of 288 patients in three equal groups

Proposed number of initial centres: two (Greifswald, Germany and Liverpool, UK).

Duration of dosing: 12 months

Treatment groups:

Group one: Two ANTOX (vers) 1.2 tablets, three times daily, Antioxidant treatment: 300 µg organic selenium, 720 mg vitamin C, 228 mg vitamin E, 2880 mg methionine per day.

Group two: Two Magnesium-L-Aspartate-hydrochloride (Magnesiocard 2,5 mmol (MGCT)) tablets, three times daily, total dose 15 mmol (365 mg) per day.

Group three: The same number of tablets as in Groups one and two but placebo instead of active drug.

Efficacy parameters:

Primary: Pain (number of days of pancreatic pain)

Secondary: Severity of pain; analgesic use for pancreatic pain; number of days of hospitalisation for conditions related to chronic pancreatitis; quality of life; markers of inflammatory response, antioxidant response, changes in urinary levels of magnesium, selenium, vitamin C and activity of the pancreatitis and pancreatic function.

Safety parameters: Toxicity; Adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have had symptoms of pancreatitis for at least one year.
2. Patients must be willing to be followed up regularly for at least one year.
3. Patients aged 5 to 75 years of age.
4. Individuals must have characteristic pancreatic pain that is either intermittent or continuous (2 or more episodes during the last 12 months)
5. Patients with documented Hereditary Pancreatitis (HP), clinically defined or proven by gene mutations in the PRSS1 Gene, or patients with Idiopathic Chronic Pancreatitis (ICP) and no mutations detected in the PRSS1 gene. This may include patients with a history of alcohol intake who have been abstinent for at least 24 month.

Exclusion Criteria:

1. Patients that do not consent to be involved in the trial, or whose parents do not consent for their children to be involved.
2. Patients or guardians of underage patients, with learning disabilities or other cognitive or sensory impairments that would prevent adequate understanding of the study requirements.
3. Patients who have had recent treatment (<3 months), or are currently receiving treatment with antioxidants or magnesium tablets.
4. Patients who have had recent (<3 months), or are currently receiving treatment with oral steroids for their pancreatic disease.
5. Patients with renal failure (serum creatinine 200 µg/l).
6. Patients with atrio-ventricular-block.
7. Serum triglyceride levels >= 1000 mg/dl.
8. Patients under the age of five years or over the age of 75 years.
9. Patients who are dependent on daily opiate analgesia (morphine or equivalent) for more than 12 months.
10. Patients who have chronic hepatic failure, or serious impairment of pulmonary, cardiac, neurological or cerebral function.
11. Patients who are participating in another drug trial.
12. Patients who are pregnant.
13. Women of childbearing age who are not using contraception.
14. Lactating mothers.
15. Any disorder that would prevent adequate absorption of the active treatment.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2005-06-06 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of days of pancreatic pain. | 1 year

SECONDARY OUTCOMES:
Disruption of activities of normal living (patient reports). | 1 year
  Number of days with limitations in activities by pancreatic pain per week, Assessment of limitation in activities by pancreatic pain (scale from 0 (no limitation) to 10 (total limitation))
Analgesic use for pancreatic pain. | 1 year
Number of days of hospitalisation for conditions related to pancreatitis. | 1 year
Quality of life (QoL) measures. | 1 year
Markers of inflammatory response and activity of the pancreas. | 1 year
Changes in urinary levels of magnesium, selenium, and vitamin C. | 1 year
Antioxidant response as measured by urinary thiobarbituric acid levels. | 1 year
Response in patients with hereditary pancreatitis and idiopathic chronic pancreatitis. | 1 year
Correlate response with gene mutations underlying hereditary pancreatitis (PRSS1, other) and idiopathic chronic pancreatitis (SPINK1, Cystic Fibrosis Transmembrane Conductance Regulator (CFTR), other). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Markus M Lerch, Professor,MD, Principal Investigator — Klinik für Innere Medizin A, Universitätsmedizin Greifswald; Julia V Mayerle, Professor,MD, Principal Investigator — Medizinische Klinik II, Klinikum der Universität München; Christopher Halloran, Professor,MD,FRCS, Principal Investigator — Molecular and Clinical Cancer Medicine, University of Liverpool

REFERENCES:
- See also: Department of Medicine A; Universitätsmedizin Greifswald — http://www.pancreas.de